CLINICAL TRIAL: NCT05689268
Title: EUS-portal Pressure Gradient (EUS-PPG). Prospective Study Compared With Hepatic Venous Pressure Gradient (HVPG)
Brief Title: EUS-PPG vs HVPG in Portal Hypertension
Acronym: GRAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General Universitario de Alicante (Other)
Responsible Party: Principal Investigator, Jose Ramon Aparicio Tormo, Head of Endoscopy Unit, Hospital General Universitario de Alicante
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PI2021-135
Record Dates: First submitted 2021-12-01; First posted 2023-01-19 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Cirrhosis; Portal Hypertension
Keywords: EUS; Endoscopic ultrasound; Portal Hypertension; Portal pressure gradient; Hepatic venous pressure gradient
MeSH Terms: conditions — Fibrosis; Hypertension, Portal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EUS-PPG and HVPG (Other): EUS-PPG and HVPG will be measured in all patients. Under deep sedation with propofol, an echoendoscopy will be performed. After identifying the left or middle suprahepatic vein, it will be punctured with a standard 22 G needle. The needle will be previously purged with heparinized saline and connected to a venous pressure monitor via an arterial pressure system, which will be calibrated to zero at the level of the axillary midline, at the level of the atrium. Subsequently, the left portal vein will be identified from the stomach or duodenum, repeating the procedure. From each vessel 3 measurements will be taken by flushing 1-2 ml of heparinized saline. The mean of the three measurements will be obtained.
  On the same day or on successive days HVPG measurement will be performed.
  Interventions: Diagnostic Test: EUS-PPG and HVPG

INTERVENTIONS:
Diagnostic Test: EUS-PPG and HVPG — EUS-PPG and HVPG will be measured in all patients. Under deep sedation with propofol, an echoendoscopy will be performed. After identifying the left or middle suprahepatic vein, it will be punctured with a standard 22 G needle. The needle will be previously purged with heparinized saline and connected to a venous pressure monitor via an arterial pressure system, which will be calibrated to zero at the level of the axillary midline, at the level of the atrium. Subsequently, the left portal vein will be identified from the stomach or duodenum, repeating the procedure. From each vessel 3 measurements will be taken by flushing 1-2 ml of heparinized saline. The mean of the three measurements will be obtained.
  On the same day or on successive days HVPG measurement will be performed.

SUMMARY:
The objective of this study is to evaluate the correlation of the calculated portal pressure gradient (PPG) obtained by direct portal and hepatic pressure measurements with a conventional 22 G needle guided by EUS and indirect portal vein pressure measurements using the interventional radiology based hepatic venous pressure gradient (HVPG) procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Undergoing evaluation for chronic liver disease or portal hypertension
* Signed informed consent

Exclusion Criteria:

* Uncorrectable coagulopathy (INR above 1.5)
* Uncorrectable thrombocytopenia (Platelets under 50,000)
* Anticoagulation or antiplatelet therapy that cannot be discontinued
* Biliary obstruction
* Grade II ascites or more
* Intrahepatic portal vein thrombosis
* Pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Intra-class correlation coefficient between portal pressure gradient measurement by EUS and hepatic venous pressure gradient measurement measured by interventional radiology. | 1 day
  Portal pressure gradient measurement will be performed by direct echoendoscopy-guided puncture with a 22 G needle of the portal vein and the suprahepatic vein. On the same day or on successive days, hepatic venous pressure gradient determination will be performed by interventional radiology. For this purpose, the free hepatic venous pressure and the wedged pressure will be measured using a balloon catheter and jugular approach, following the usual procedure.

SECONDARY OUTCOMES:
Technical success of both procedures measured as the number of procedures successfully performed divided by the total number of patients. | 1 day
  The percentage of echoendoscopy-guided portal pressure gradient (EUS-PPG) measurements versus the percentage of successful hepatic venous pressure gradient (HVPG) measurements using Chi-square will be compared.
Adverse effects at 30 days after each procedure by clinical follow-up of patients at 24 hours, 7 days, and 30 days using the American Society of Gastrointestinal Endoscopy Severity grading system, from mild to fatal. | 30 days
  Proportion of adverse events in the EUS-PPG and HVPG using Chi-square.

CONTACTS AND LOCATIONS:
Locations (1):
- Unidad de Endoscopia. Hospital General Universitario de Alicante, Alicante, Spain